CLINICAL TRIAL: NCT02952651
Title: Prediction of Fluid Responsiveness Using Respiratory Variation in Pulse Oximeter Plethysmography in Children Undergoing Major Surgery
Brief Title: Prediction of Fluid Responsiveness in Children Undergoing Major Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H1609-066-791
Record Dates: First submitted 2016-10-19; First posted 2016-11-02 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Hypovolemia
MeSH Terms: conditions — Hypovolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children with hypovolemic state (Experimental): Pulse oximeter plethysmography (POP) waveforms are obtained for 90 seconds in children with hypovolemic signs including hypotension, decreased urine output and central venous pressure less than 5 mmHg. Then, intravenous crystalloid fluid 10 mL/kg is infused for 15 min. Delta POP is calculated, and diagnostic power of delta POP for fluid responsiveness will be evaluated.
  Interventions: Procedure: Pulse oximeter

INTERVENTIONS:
Procedure: Pulse oximeter — When there are clinical signs of hypovolemia, such as hypotension, decreased urine output and central venous pressure less than 5 mmHg, POP waveforms are obtained from each index finger, which pulse oximeter sensor is applied by increasing contact force (from 0 to 1.4N, being increased by 0.2-0.3N). Then intravenous crystalloid 10 mL/kg is infused for 15 min.

SUMMARY:
The purpose of this study is to evaluate predictability of a respiratory variation in pulse oximeter plethysmography for fluid responsiveness in children undergoing major surgery.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate predictability of a a respiratory variation in pulse oximeter plethysmography (delta POP) for fluid responsiveness in children undergoing major surgery.

When there are clinical signs of hypovolemia, such as hypotension, decreased urine output and central venous pressure less than 5 mmHg, the study will be started. At index fingers of both hand, pulse oximeter sensors are applied by gradually increasing the contact force (from 0 to 1.4N, being increased by 0.2-0.3N). Then, pulse oximeter plethysmography (POP) waveforms are obtained for 90 seconds. Then, intravenous crystalloid fluid 10 mL/kg is infused for 15 min.

To evaluate the change of cardiac output, transesophageal or transthoracic echocardiography is performed before and after fluid administration. In addition, hemodynamic parameters including pulse pressure variation, systolic pressure variation, pleth variability index and central venous pressure are also recorded before and after fluid administration.

Finally, patients will be divided into fluid responder group and non-responder group. If stroke volume index measured using echocardiography increases over 15% after fluid administration, the patient will be fluid responder.

Delta POP (%) obtained from each finger with different contact force is calculated as follows;(POPmax - POPmin)/{(POPmax + POPmin)/2}. Using receiver operating characteristic curve, diagnostic power of delta POPs from different contact forces for fluid responsiveness will be evaluated. In addition, difference between delta POP from low contact force and that from high contact force will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

- Children who will be scheduled for major surgery requiring invasive hemodynamic monitoring

Exclusion Criteria:

* renal, hepatic and pulmonary disease
* preoperative infection: increased C-reactive protein, whith blood cell count over 10,000, and with fever
* genetic and hematologic disease
* ventricular dysfunction
* increased intracranial pressure

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2018-01-20 (Actual); Study Completion 2018-01-20 (Actual)

PRIMARY OUTCOMES:
The ability of delta POP for prediction of fluid responsiveness in children | Before and after fluid administration (total 20 min)
  Delta POP (%) obtained from each finger with different contact force is calculated as follows;(POPmax - POPmin)/{(POPmax + POPmin)/2}. Delta POP differs according to contact force. After calculation of each delta POP, we will evaluate the ability to predict fluid responsiveness of delta POP using receiver operating characteristic curve.

CONTACTS AND LOCATIONS:
Locations (1):
- SNUH, Seoul, Jongro Gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided